CLINICAL TRIAL: NCT04677049
Title: A Phase I-II Study of Niacin in Patients With Newly Diagnosed Glioblastoma Receiving Concurrent Radiotherapy and Temozolomide Followed by Monthly Temozolomide
Brief Title: Study of Niacin in Glioblastoma
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment has been placed on hold to determine evaluability of currently enrolled patients. Recruitment will remain on hold until evaluability is confirmed. If fewer than 48 evaluable patients are achieved, the study will be re-opened to accrual.
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NiacinCNS2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma IDH (Isocitrate Dehydrogenase) Wildtype
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Niacin; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niacin (Experimental): Niacin controlled release technology (CRT):
  Niacin CRT™ is to be started 7 days before concurrent Radiation Therapy (RT)- Temozolomide (TMZ) treatment.
  Chemo/Radiation Therapy:
  For all patients, regardless of the phase of the study, concurrent RT and TMZ for 6 weeks followed by 6-12 cycles of monthly TMZ will be given.
  Concurrent Temozolomide:
  TMZ will be administered from the first to the last day of RT at 75 mg/m2 orally (PO) for a maximum of 49 days.
  Monthly Temozolomide:
  Cycles of chemotherapy Day 1 to Day 5 every 28 days will start 28 days (+/- 2 days) after the end of RT-TMZ. First cycle of TMZ is administered at 150 mg/m2 Day 1-Day 5 by mouth (PO) and increased to 200 mg/m2 Day 1-Day 5 PO from cycle 2 onwards if well tolerated. While 6 cycles are standard of care, the Neuro-Oncologist may continue up to 12 cycles if clinically appropriate.
  Interventions: Drug: Niacin CRT

INTERVENTIONS:
Drug: Niacin CRT — A controlled release technology (CRT) tablet of Niacin
  Other Names: Nicotinic acid; Vitamin B3

SUMMARY:
This is a single institution Phase I-II study to evaluate the tolerability and Maximum Tolerated Dose (MTD) (Phase I) and efficacy (Phase II) of adding Niacin CRT™ to standard first line treatment (concurrent Radiation Therapy (RT) and Temozolomide (TMZ) following by monthly TMZ - AKA Stupp protocol) in patients with newly diagnosed glioblastoma isocitrate dehydrogenase (IDH) wild type.

DETAILED DESCRIPTION:
During the Phase I stage Niacin CRT™ dose will be escalated every 4 weeks until the maximum tolerated dose (MTD) is determined. The MTD dose will be prescribed to patients during the Phase II stage.

During the Phase I study a sample of blood at baseline, at each level dose of Niacin CRT™, and every two months during the maintenance phase while on Niacin CRTTM will be sent to a lab to evaluate the peripheral activity of Niacin CRT™ in innate immune system cells. These samples will be taken at the time of routine standard of care lab work.

Based on prior clinical trials evaluating niacin extended release formulation for the management of dyslipidaemias there is vast experience on dose escalation of niacin. One of the main side effects is flushing that is ameliorated by escalating doses in intervals no shorter than 4 weeks and usually decreases with time.

Following this schema, there is no increase in dose coinciding with TMZ while administered in a 5/28 days schedule (given daily for 5 days of each 28-day cycle). This will not only improve tolerance but also will allow us to differentiate potential adverse events from chemotherapy from the ones from Niacin CRT™.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years old to 75 years old inclusive.
* New diagnoses of glioblastoma IDH wild type.
* ECOG 0-2 (Appendix I).
* Candidates for concurrent standard first line treatment according to their Neuro-Oncologist and Radiotherapy Oncologist after maximal safe debulking neurosurgery. Patients that only had biopsy are included as long as pathology confirms the diagnoses and it is considered the maximal safe procedure for that patient.
* Adequate hematological, renal and hepatic function (see details in Section 4.1 of the protocol).
* Absence of known human immunodeficiency virus (HIV) infection, chronic hepatitis B or hepatitis C infection.
* Absence of any other serious medical condition according to the medical judgment of the Qualified Investigator prior to registration.
* Absence of any medical condition, which could interfere with oral medication intake.
* Signed informed consent.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Glioblastoma, IDH-mutant.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years. Additionally, any low grade or low risk malignancy not requiring treatment will not exclude a patient from participation in the trial.
* Known hypersensitivity to niacin.
* Inability to provide informed consent.
* Active liver disease or unexplained persistent elevations of serum transaminases.
* Active peptic ulcer or active gastrointestinal bleeding.
* Unstable angina or myocardial infarction within 6 months.
* Symptomatic gout.
* Patients on 3-hydroxy-3-methylglutaryl-coenzyme (HMG-COA reductase) inhibitors that cannot discontinue them at least 2 weeks before starting Niacin CRT™.
* Any prior systemic treatment for glioblastoma (standard, evidence based or experimental) or radiotherapy/radiosurgery.
* Individuals with MRI non-compatible metal in the body, or unable to undergo MRI procedures including allergy to gadolinium.
* Patients unfit for any treatment component, including contraindications for radiotherapy or Connective Tissue Disease.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has known psychiatric or substance abuse disorders that would interfere with compliance with the requirements of the trial.
* Pregnant, breast-feeding, unable and/or unwilling to use contraception methods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining the Maximum Tolerated Dose | Up to 24 weeks after registration onto the study
  To evaluate and determine maximum tolerated dose (MTD) of Niacin CRT added to concurrent radiotherapy (RT) and temozolomide (TMZ) in patients with newly diagnosed glioblastoma (GB).
Evaluating if Niacin CRT Improves Glioblastoma Survival Rates | 6 months after determining the maximum tolerated dose which can last up to 24 weeks after registration onto the study
  To evaluate if adding Niacin CRT to current standard first line treatment of GB improves progression free survival (PFS) at 6 months.

SECONDARY OUTCOMES:
Effect of Niacin CRT in Peripheral Monocytes | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To evaluate the effect of Niacin CRT in peripheral monocytes by comparing control monocytoid cells to those that have been treated with Niacin.
Response Rate Associated with Niacin | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To determine the response rate associated with the investigational regimen.
Overall Survival Rate Associated with Niacin | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To determine the overall survival (OS) associated with the investigational regimen.
Quality of Life While on Study using EORTC QLQ-C30 Questionnaires | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To determine Quality of Life (QOL) that will be evaluated throughout the study using EORTC QLQ-C30 questionnaires.
Quality of Life While on Study using EORTC BN-20 Questionnaires | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To determine Quality of Life (QOL) that will be evaluated throughout the study using EORTC BN-20 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Roldan Urgoiti, MD, Principal Investigator — Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre
Locations (1):
- Tom Baker Cancer Centre/Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poon CC, Hagen KM, Sarkar S, Mirzaei R, Silva C, Ueno A, de Robles P, Roldan-Urgoiti G, Yong VW. Niacin Modulates Immune Responses in a Phase I Dose-Escalation Clinical Trial of Newly Diagnosed Glioblastoma. Neurol Neuroimmunol Neuroinflamm. 2026 Mar;13(2):e200530. doi: 10.1212/NXI.0000000000200530. Epub 2026 Feb 3. PMID 41632924